CLINICAL TRIAL: NCT05052866
Title: Development of Ryan Companion Robot for Assisting Elderly People With Alzheimer's Disease
Brief Title: Ryan Companion Robot for Assisting Elderly People With Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DreamFace Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-02
Record Dates: First submitted 2021-09-04; First posted 2021-09-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Alzheimer Disease, Early Onset
MeSH Terms: conditions — Alzheimer Disease | interventions — Robotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot Intervetnion (Experimental): Participants in this Arm will interact with Ryan Companionbot.
  Interventions: Behavioral: Social Robot

INTERVENTIONS:
Behavioral: Social Robot — Participants will interact with a social robot companionbot for a period of 8-10 weeks. The robot will stay in participants' apartments.

SUMMARY:
The objective of this project is to conduct research and a pilot study to demonstrate the potential clinical impact and technical feasibility of a socially-assistive robot, called Ryan Companionbot (hereafter Ryan), for life improvement and intervention of persons with early stage Alzheimer's disease (AD) and AD related dementia (ADRD). Earlier phases of this project demonstrated the feasibility and scalability of using emotion recognition technology based on cutting-edge natural language processing and artificial intelligence technologies to improve mood and lessen depression symptoms of persons with early stage AD/ADRD. In this phase, the investigators will utilize an aesthetically pleasing updated Ryan (V2.0) with emotion recognition and natural language processing for enhanced conversations to address the needs of the individuals with AD/ADRD and their healthcare providers as well as to test the effectiveness of Ryan by comparing participants pre- and post-treatment by analyzing several blood biomarkers related to AD/ADRD and depression. The investigators will recruit thirty participants from local senior living facilities based on their cognitive performance as assessed by the Saint Louis University Mental Status (SLUMS) score. SLUMS is commonly used as a simple screening/assessment test in senior living facilities. As part of the recruitment, the investigators will show prospective participants a video recording of a previous senior volunteer interacting with Ryan to give new recruits an idea of the socially assistive robot technology.

ELIGIBILITY:
Inclusion Criteria:

* HAVING EARLY STAGE AD/ADRD AS ASSESSED BY THE SLUMS SCORE (BETWEEN 15-26),
* VERBAL SKILL TO INTERACT,
* BEING AVAILABLE FOR A PERIOD OF 8-10 WEEKS TO INTERACT WITH RYAN,
* HEALTHY INDIVIDUALS WEIGHING AT LEAST 110 POUNDS (FOR SAFE COLLECTION OF BLOOD SAMPLES).

Exclusion Criteria:

* AGGRESSIVE BEHAVIOR
* DIAGNOSTICS OF SEVERE DEMENTIA OR MEMORY LOSS
* ACUTE PHYSICAL ILLNESS THAT IMPAIRS ABILITY TO PARTICIPATE
* DURING THE STUDY IF A PARTICIPANT'S MID-STUDY SLUMS SCORE IS LESS THAN 15 (INDICATING MORE SEVERE DEMENTIA) AND/OR THE PHQ-9 IS EQUAL TO OR GREATER THAN 20, THE CUTOFF FOR SEVERE DEPRESSION, THE RESEARCHERS WILL REMOVE THE PARTICIPANT FROM THE STUDY
* IF A PERSON IS UNCOMFORTABLE WITH BLOOD DRAW, HE/SHE IS EXCLUDED FROM THE STUDY.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Robot Usage Time | 8-10 weeks
  How much time the user spends with the robot
Conversation Time | 8-10 weeks
  How much time the user spends in conversation with the robot
Facial Expression | 8-10 weeks
  Facial expressions throughout conversation with robot
Sentiment Analysis | 8-10 weeks
  Speech is analyzed and is either classified as positive, neutral, or negative.
Amyloid-Beta - Alzheimer's disease | 8-10 weeks" Blood will be collected once before the robot is dropped off, once during the midpoint of the study, and once at the end of the study.
  Levels of Amyloid-beta will be analyzed from blood collected at time of study. Amyloid-beta peptide is believed to drive Alzheimer's disease pathogenesis and is the main component of amyloid plaques.
Phospho-Tau - Alzheimer's disease | 8-10 weeks" Blood will be collected once before the robot is dropped off, once during the midpoint of the study, and once at the end of the study.
  Levels of Phospho-tau will be analyzed from blood collected at time of study. In Alzheimer's disease, tau instead of stabilizing microtubules detach from them and form tangles in the neurons.
brain derived neurotrophic factor (BDNF) - depression | 8-10 weeks" Blood will be collected once before the robot is dropped off, once during the midpoint of the study, and once at the end of the study.
  Levels of BDNF will be analyzed from blood collected at time of study. BDNF is believed to be decreased in patients experiencing depression.
serotonin (5-HT) - this is for depression | 8-10 weeks" Blood will be collected once before the robot is dropped off, once during the midpoint of the study, and once at the end of the study.
  Levels of Serotonin will be analyzed from blood collected at time of study. Serotonin is a neurotransmitter that has been linked to depression when depleted.

SECONDARY OUTCOMES:
SLUMS score | The Saint Louis University Mental Status exam will be administered three times during the 8-10 week period. It is a 11 set questionnaire that is scored between 1 and 30 points. A higher score is a better outcome.
  The SLUMS test is a screening tool for dementia and mild cognitive impairment.
PHQ-9 | The Patient Health Questionnaire-9 will be administered three times during the 8-10 week period. The score is between 0 and 27. Each questions is scored between "0" (not at all) to "3" (nearly every day). A higher score is a worse outcome.
  The Patient Health Questionnaire-9 is a major depressive disorder screening module.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Melgar, BS, Study Director — University of Denver/ DFT
Locations (1):
- Eaton Senior Communities, Lakewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will share the final results and the data with other researchers after the data collection is over.